CLINICAL TRIAL: NCT00522210
Title: A Comparison of Insulin Detemir in a BID Insulin Regimen Versus a TID Insulin Regimen in Children With Type 1 Diabetes: A Randomized Controlled Trial
Brief Title: Comparison of a Twice Daily Versus a Three Times Daily Insulin Regimen in Children With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Josephine Ho, Pediatric Endocrinologist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-20635
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2011-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; children; long acting insulin analogue; hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Isophane Insulin, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BID insulin with LA analogue (Experimental): Treatment Group: BID Insulin Regimen with Long Acting Insulin Analogue (Detemir)
  Interventions: Drug: Detemir
- Standard TID insulin (Active Comparator): Active Control Group: Usual TID Insulin Regimen (intermediate insulin- Humulin N or Novolin NPH)
  Interventions: Other: Novolin NPH or Humulin N

INTERVENTIONS:
Drug: Detemir — Patients will discontinue their usual bedtime dose of intermediate acting insulin and replace this with the same unit dose of detemir at supper time. The detemir will not be mixed with the rapid acting insulin and will be given as a separate injection. The patient's morning dose of intermediate acting insulin will be decreased by 20% to adjust for the longer duration of action of detemir. Doses of rapid acting insulin will remain the same at breakfast and at supper.
  Other Names: Levemir
  Arms: BID insulin with LA analogue
Other: Novolin NPH or Humulin N — Patients will continue on their usual insulin regimen of insulin three times per day. Intermediate and rapid acting insulin at breakfast, rapid acting insulin at supper, and intermediate acting insulin at bedtime.
  Arms: Standard TID insulin

SUMMARY:
The purpose of this study is to determine whether there is a difference in blood sugar control (as measured by hemoglobin A1c (HA1c)), in children given twice daily insulin injections incorporating a new long acting insulin analogue (detemir) compared to children using their current three times a day insulin injections (with intermediate and rapid acting insulin).

DETAILED DESCRIPTION:
Children with type 1 diabetes (DM1) can only be treated with subcutaneous insulin at the present time in Canada. It has been shown that intensive insulin treatment using at least three times daily (TID) insulin injections achieves superior blood glucose control with less long term complications of diabetes than conventional insulin treatment using once daily (OD) or twice daily (BID) insulin injections. However, many patients find it difficult to adhere to TID insulin injections since it is an invasive and painful therapy, which results in frequent insulin omission.

This study is a randomized controlled open-labeled non-inferiority trial to compare the glycemic control as measured by HbA1c after 6 months of a BID insulin regimen using detemir insulin, or the currently used TID insulin with intermediate acting insulin (Novolin NPH or Humulin N). Patients will be randomized to either the active control group (standard TID regimen) or the treatment group (BID regimen with new long acting insulin analogue). A run-in period of 1 month will be used to facilitate the change in insulin regimen. Insulin doses will be adjusted by weekly phone contact with the research nurse for one month prior to baseline blood work. Patients will continue on the same diet and exercise routine as recommended by their usual diabetes team. They will also be seen every 3 months by the research nurse to review blood glucose, assess height and weight and arrange for blood work to be done in conjunction with their routine bloodwork. All patients will continue to be seen by their usual diabetologist, nurse, and dietician at their regularly scheduled clinic visits (every 3 months).

Outcomes include: HA1c between groups at 6 months (surrogate marker of metabolic control for diabetes measured through a venous or capillary blood sample), frequency of adverse events (severe hypoglycemia, mild hypoglycemia, episodes of diabetic ketoacidosis, weight gain), diabetes quality of life for youth (DQOL).

ELIGIBILITY:
Inclusion Criteria:

1. Children with DM1 6-17 years old that are currently on a TID regimen of insulin with rapid acting insulin and intermediate acting insulin.
2. Currently being followed at the Alberta Children's Hospital Diabetes Clinic.
3. Duration of diabetes of at least 12 months.

Exclusion Criteria:

1. Children younger than 6 years of age will be excluded since long-acting analogue has not been approved in children younger than 6 years old.
2. Children with compromised metabolic control (HA1c greater than 10%).
3. Children with other chronic underlying medical conditions that could affect glycemic control i.e. uncontrolled hypothyroidism, hyperthyroidism, celiac disease, etc.
4. Language or psychosocial barrier preventing the family from completing the study.
5. Diabetes duration of less than 12 months.
6. Participation in other clinical trials with specified clinic visit schedule.
7. Patients currently on insulin pump therapy or multiple daily injections of greater than three injections per day.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C | 6 months

SECONDARY OUTCOMES:
Number of episodes of hypoglycemia (severe and mild) | 6 months
Number of episodes of diabetic ketoacidosis (DKA) | 6 months
Body Mass Index (BMI) kg/m2 | 6 months
Diabetes Quality of Life Questionaire-youth version | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Ho, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

REFERENCES:
- [Result] Ho J, Huang C, Nettel-Aguirre A, Pacaud D. Insulin detemir in a twice daily insulin regimen versus a three times daily insulin regimen in the treatment of type 1 diabetes in children: A pilot randomized controlled trial. Int J Pediatr Endocrinol. 2011 Nov 8;2011(1):15. doi: 10.1186/1687-9856-2011-15. PMID 22067102